CLINICAL TRIAL: NCT05403918
Title: Effects of Conventional Physical Therapy With and Without Scapular Stabilization Exercises on Pain, Function, Scapular Dyskinesia and Proprioception in Patients With Adhesive Capsulitis.
Brief Title: Effects of Conventional Physical Therapy With and Without Scapular Stabilization Exercises in Adhesive Capsulitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0119
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; scapular dyskinesis; proprioception; scapular stabilization exercises
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physiotherapy (Active Comparator): 15 patients will receive conventional physiotherapy including a hot pack, TENS, therapeutic ultrasound, shoulder anteroposterior, posteroanterior, and inferior glides followed by active and active-assisted range of motion exercises, isometric exercises, Codman's pendulum exercises, wand, pulley, and finger ladder exercises.
  Interventions: Other: conventional physiotherapy
- scapular stabilization exercises along with conventional physiotherapy (Experimental): 15 participants will receive conventional treatment along with scapular stabilization exercises program consisting of strengthening exercises (Middle Trapezius, Lower Trapezius, Serratus Anterior, and Rhomboid Muscles) and stretching exercises (Pectoralis Minor, Levator Scapulae, Upper Trapezius, Teres Major). Appropriate exercises will be given to patients according to the type of Scapular Dyskinesia.
  Interventions: Other: scapular stabilization exercises along with conventional physiotherapy

INTERVENTIONS:
Other: conventional physiotherapy — Hot pack, TENS, and therapeutic ultrasound will be applied for 10 minutes. Then glides will be given 30 x 3 times in grades III and IV. The rest of the exercises will be prescribed as 3 sets for 10 repetitions with 2 minutes of rest between sets for 6 weeks with respect to 3 sessions per week.
  Arms: conventional physiotherapy
Other: scapular stabilization exercises along with conventional physiotherapy — Each stretch will be repeated 3 times. Each active exercise will be progressed from 3 sets of 10 reps to 3 sets of 15 reps. If the subject easily completed 3 sets of 15 reps of active exercise, they will go on to resisted exercises. These will be performed once a day, for 6 weeks, 3 sessions per week.
  Arms: scapular stabilization exercises along with conventional physiotherapy

SUMMARY:
The objective of this study will be to determine the Effects of conventional physical therapy with and without scapular stabilization exercises on pain, function, scapular dyskinesia, and proprioception in patients with adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis is characterized by the gradual onset of severe shoulder pain with the progressive limitation of active and passive glenohumeral range of motion. Due to capsular tightness and pain, scapular positioning and proprioception get affected. An increase in the abnormal positioning of the scapula and proprioception deficit disturbs the whole biomechanics of the shoulder joint and are the main causes of residual pain and stiffness following PT treatment.

In previous studies, several studies have reported the effects of scapular stabilization exercises on pain, ROM, and function but there is a paucity of literature available on specifically addressing scapular dyskinesis and joint position sense in patients with adhesive capsulitis. Scapular stabilization techniques will help to improve proprioception and the length-tension relationship of the scapular muscles, which may effectively reduce the time taken for the rehabilitation of the patient with adhesive capsulitis of the shoulder joint.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic adhesive capsulitis for more than 4 months (Stage 2)
* Unilateral idiopathic adhesive capsulitis
* Shoulder Pain on NPRS ≥5
* Restricted ROM (loss of ≥ 25% relative to non-involved shoulder in one or multidirectional)
* Patients volunteered to participate in the study and signed informed consent.

Exclusion Criteria:

* History of shoulder surgery or manipulation under anesthesia
* Unstable fractures, rheumatoid arthritis and those with severe joint pain unrelieved by rest
* Neurologic deficits affecting shoulder functioning during daily activities
* Pain or disorders of the cervical spine, elbow, wrist, or hand
* Other pathological conditions involving the shoulder (rotator cuff tear, tendinitis, etc.)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
NPRS for pain | 6th week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Bubble inclinometer for shoulder ROM and JPS | 6th week
  A bubble Inclinometer is used for measuring the range of motion and joint position sense in patients.
SPADI for pain and disability | 6th week
  Shoulder pain and disability index include thirteen questions measuring pain and disability on an eleven-point scale. O being no pain, difficulty and 10 being worst pain and difficulty.
LSST for static scapular movement | 6th week
  A lateral scapular slide test is used to assess scapular position in shoulder pathologies.
SDT for dynamic scapular movement | 6th week
  The scapular dyskinesia test is used to measure dynamic scapular movement.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Physical therapy department, Qari Hospital, Okara., Okara, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gulwani AH. A study to find out the effect of scapular stabilization exercises on shoulder ROM and functional outcome in diabetic patients with stage 2 adhesive capsulitis of the shoulder joint - An interventional study. International Journal of Science and Healthcare Research. 2021;Vol.5(Issue: 2).
- [Background] Rajpurohit B, Anap D. Scapular dyskinesis among patients with shoulder dysfunction-A Cross Sectional Study. VIMS JOURNAL OF PHYSICAL THERAPY. 2021;3(1).
- [Background] Panagiotopoulos AC, Crowther IM. Scapular Dyskinesia, the forgotten culprit of shoulder pain and how to rehabilitate. SICOT J. 2019;5:29. doi: 10.1051/sicotj/2019029. Epub 2019 Aug 20. PMID 31430250
- [Background] Ager AL, Borms D, Bernaert M, Brusselle V, Claessens M, Roy JS, Cools A. Can a Conservative Rehabilitation Strategy Improve Shoulder Proprioception? A Systematic Review. J Sport Rehabil. 2020 Jul 31;30(1):136-151. doi: 10.1123/jsr.2019-0400. PMID 32736342
- [Background] Bhale AA, Wani SK. Evaluation of shoulder kinesthesia in patients with unilateral frozen shoulder. 2019.
- [Background] Turgut E, Duzgun I, Baltaci G. Effects of Scapular Stabilization Exercise Training on Scapular Kinematics, Disability, and Pain in Subacromial Impingement: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Oct;98(10):1915-1923.e3. doi: 10.1016/j.apmr.2017.05.023. Epub 2017 Jun 24. PMID 28652066
- [Background] Tang L, Chen K, Ma Y, Huang L, Liang J, Ma Y. Scapular stabilization exercise based on the type of scapular dyskinesis versus traditional rehabilitation training in the treatment of periarthritis of the shoulder: study protocol for a randomized controlled trial. Trials. 2021 Oct 18;22(1):713. doi: 10.1186/s13063-021-05654-2. PMID 34663424
- [Background] Kim JT, Kim SY, Oh DW. An 8-week scapular stabilization exercise program in an elite archer with scapular dyskinesis presenting joint noise: A case report with one-year follow-up. Physiother Theory Pract. 2019 Feb;35(2):183-189. doi: 10.1080/09593985.2018.1442538. Epub 2018 Feb 26. PMID 29482465
- [Background] Nodehi Moghadam A, Rahnama L, Noorizadeh Dehkordi S, Abdollahi S. Exercise therapy may affect scapular position and motion in individuals with scapular dyskinesis: a systematic review of clinical trials. J Shoulder Elbow Surg. 2020 Jan;29(1):e29-e36. doi: 10.1016/j.jse.2019.05.037. Epub 2019 Aug 13. PMID 31420226
- [Background] Krantz R, Rasmussen-Barr E. The Swedish version of the Lumbar Spine Instability Questionnaire: A clinimetric study of validity and reliability. Physiother Theory Pract. 2023 Jan;39(1):154-162. doi: 10.1080/09593985.2021.1999353. Epub 2021 Nov 1. PMID 34724863
- [Background] Shadmehr A, Sarafraz H, Heidari Blooki M, Jalaie SH, Morais N. Reliability, agreement, and diagnostic accuracy of the Modified Lateral Scapular Slide test. Man Ther. 2016 Aug;24:18-24. doi: 10.1016/j.math.2016.04.004. Epub 2016 Apr 19. PMID 27317502
- [Background] Christiansen DH, Moller AD, Vestergaard JM, Mose S, Maribo T. The scapular dyskinesis test: Reliability, agreement, and predictive value in patients with subacromial impingement syndrome. J Hand Ther. 2017 Apr-Jun;30(2):208-213. doi: 10.1016/j.jht.2017.04.002. Epub 2017 May 29. PMID 28571725